CLINICAL TRIAL: NCT03711045
Title: An Eye Tracking Study of Affective Disorder Patients With Suicide Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Lingjiang Li, President of Chinese Psychiatry Society of Chinese Medical Association, Central South University
Other Study IDs: Second Xiangya hospital CSU; Mental Health Insititute (Other: Second Xiangya Hospital)
Record Dates: First submitted 2018-10-11; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Suicide
Keywords: eye-tracking; eye movement; saccade
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suicide Risk Group: patients with affective disorders(eg. bipolar disorder, major depression disorder) also have a history of suicide attempt in the past 6 months.
  Interventions: Behavioral: eye-tracking
- Disorder Control Group: patients with affective disorders(eg. bipolar disorder, major depression disorder) and without suicide ideation or behavior.
  Interventions: Behavioral: eye-tracking
- Healthy Control Group
  Interventions: Behavioral: eye-tracking

INTERVENTIONS:
Behavioral: eye-tracking — After completing a demographics form, theBeck Depression Inventory,Beck Anxiety Inventory,Barratt Impulsiveness Scale and Ruminative Response Scale-21, each participant has to go to the eye-tracking room and seats in a height adjustable chair and places their chin in a chin rest which was positioned to make sure all participants' eye are in the same location relative to the camera and the monitor.
  There are 18 trials and 2 filler trials in the free-view task, each of which contains 4 pictures on the same screen for 25 seconds. There is also a gap screen between each trial lasting for 2 seconds when participants were asked to fixate in the center of the screen. During the experiment, participants are instructed to watch the screen as naturally as possible, and the initial location of the fixation of each trial and the total dwell time of each emotional images(negative, happy, neutral and suicide-related)and the changes of the pupil size were recorded.

SUMMARY:
This research tries to investigate the validity and reliability of eye-tracking technologies by using different paradigms (eg. free-view, pro-saccade and anti-saccade) which served as a novel way of evaluating suicide risk among affective disorder patients including bipolar and unipolar depression. All the participants including health control will be assessed by clinical interviewing, self-report assessment, cognitive evaluation and eye-tracking task.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual,DSM-IV diagnosis of depression or Bipolar disorder
* BDI-II>20(Suicide and disorder control group); BDI-II<13，no history of depression(Health control)
* Informed consent
* suicide attempt in the past 6 months(suicide risk group)

Exclusion Criteria:

* Current or past substance abuse, psychotic disorder,obsessive compulsive disorder , Post-Traumatic Stress Disorder, in the past 6 months
* History of epilepsy or head trauma
* Eye disorders
* History of electroconvulsive therapy in the past 4 weeks.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants were recruited from outpatients in psychiatric clinic and clinical psychological clinic, and inpatients residing in the mental health hospital.
  Most of the healthy volunteers were recruited from the advertisement posters in community and medical college.
  There are two steps for screening. Firstly, each person was asked to complete the BDI (Beck Depression Inventory,21-items) to evaluate the depressive symptoms. Individuals with scores less than 13 and more than 20 were enrolled for this study.
  Secondly, each individual has to be taken for a structural diagnostic interview (MINI-International Neuropsychiatric Interview, M.I.N.I.6.0.) in order to diagnosis current disorder and evaluate suicide risk by a psychiatrist who had already clinical consistency training.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
eye movement performance during free-view task | 1 hour
  The first fixated location and latency(msec)of eah trial, the total dwell time(msec) in each interest areas(IAs) during the whole trial to assess the attentional bias in the experiment.

SECONDARY OUTCOMES:
Scores in self-report assessment:Beck Depression Inventory | 5 minutes
  This scale is aimed to assess the clinical depressive symptom in the recent 7 days.
Scores in self-report assessment:Beck Anxiety Inventory | 5 minutes
  This scale is aimed to assess the clinical anxieous symptom in the recent 7 days
Scores in self-report assessment:Barratt Impulsiveness Scale | 5 minutes
  This scale is aimed to assess participant's impulsive trait.
Scores in self-report assessment:Ruminative Response Scale | 5 minutes
  This scale is aimed to assess participant's ruminative thinking process.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute & Faculty of Psychiatry of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No